CLINICAL TRIAL: NCT04981912
Title: Rituximab and High-Dose Methylprednisolone Debulking Prior to Venetoclax for Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Rituximab + High-Dose Methylprednisolone Debulking Prior to Venetoclax for CLL & SLL Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Michael Choi, Principal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 182029
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): HDMP + rituximab as a means of debulking prior to initiating venetoclax.
  Interventions: Drug: HDMP + rituximab as a means of debulking prior to initiating venetoclax.

INTERVENTIONS:
Drug: HDMP + rituximab as a means of debulking prior to initiating venetoclax. — * Patients will receive HDMP + Rituximab for 1 cycle, followed by reassessment of Tumor Burden,
  * If Tumor Burden classification is low after HDMP + Rituximab (lymph nodes < 5cm in diameter AND absolute lymphocyte count < 25k/uL), patients will initiate venetoclax dose ramp-up, with ramp-up schedule according to venetoclax package insert.
  * Patients who still have a disease burden (lymphadenopathy > 5 cm or ALC > 25k/iL) that meets criteria for medium or high risk of TLS after 1 cycle of HDMP + Rituximab are given the option to repeat a 2nd cycle of HDMP + Rituximab prior to venetoclax dose ramp-up.
  Other Names: Methylnaphthidate + Riabni/Rituxan/Ruxience/Truxima

SUMMARY:
The purpose of the study is to investigate whether the combination of rituximab and high dose methylprednisolone can be given together, can reduce the amount of cancer cells that are present prior to starting venetoclax, and therefore make it safer to take venetoclax. Patients with relapsed or refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) will be treated in this study. Subjects will be assessed for their risk of tumor lysis syndrome (TLS), a potentially serious side effect associated with venetoclax and rituxan. TLS is caused by the fast breakdown of cancer cells. TLS can lead to kidney failure or abnormal heart rhythm. Depending on their TLS risk, patients will be assigned to one of two treatment arms. Patients who are at high risk for TLS at baseline will receive HDMP/Rituximab for 1 cycle before beginning venetoclax. Patients who are at low risk for TLS at baseline will not receive HDMP/Rituximab and will instead start directly with venetoclax. Once the proper dose of venetoclax is reached, both arms will continue venetoclax for up to 2 years and receive rituximab for 5 cycles. The purpose is to determine if HDMP/Rituximab prior to venetoclax is efficient at reducing tumor burden and lowering the risk of developing TLS. Although all of these drugs are approved by the FDA for the treatment of patients with CLL or SLL, and although the combination of rituximab and venetoclax is approved by the FDA for the treatment of patients with CLL or SLL, the combination and dosing schedule in this trial are considered experimental.

DETAILED DESCRIPTION:
Objectives:

Primary:

1. To determine the percentage of patients who have a reduction of lymphadenopathy (from greater than to less than 5 cm in largest diameter) and/or absolute lymphocyte count (from greater than to less than 25k/uL) following 1 or 2 cycles of HDMP + rituximab.

Secondary:

1. To determine the rate of laboratory or clinical TLS with this strategy.
2. To determine the safety (CTCAE4) of this approach.
3. To determine the overall efficacy (iwCLL) of this overall strategy.
4. To determine the percentage of patients who have undetectable minimal residual disease in the bone marrow.

Endpoints:

Primary:

1. Percentage of patients that have a decrease in tumor burden from levels of disease that meet "Medium/High-tumor burden" criteria to meet "Low tumor burden" criteria for disease burden following 1 or 2 cycles of HDMP + Rituximab.

Secondary:

1. Percentage of patients that have a decrease in tumor burden from levels of disease that meet "Medium/High-tumor burden" c criteria to meet "Low tumor burden" criteria for disease burden following 1 cycle of HDMP + Rituximab.
2. Percentage of patients that have a decrease in tumor burden from levels of disease that meet "Medium/High-tumor burden" criteria to meet "Low tumor burden" criteria for disease burden following 2 cycles of HDMP + Rituximab.
3. Rate of laboratory TLS (from start of treatment until completion of venetoclax ramp-up)
4. Rate of clinical TLS (from start of treatment until completion of venetoclax ramp-up)
5. Adverse events by CTCAE4 definitions
6. Overall Response rate, Partial Response rate, and Complete response rate per iwCLL criteria after 9 months of venetoclax and at completion of treatment.
7. Undetectable minimal residual disease (MRD) rate based on bone marrow biopsy after 9 months of venetoclax, and at completion of treatment.

Single center, open-label, pilot/feasibility study to determine the feasibility of HDMP/R as a debulking approach prior to venetoclax.

Patients with CLL/SLL who require therapy, and have disease burden meeting criteria for Medium or High Risk Tumor Burden (based on: lymph nodes >/= 5 cm in diameter and/or absolute lymphocyte count >/= 25k/uL) are enrolled.

* Patients will receive HDMP + Rituximab for 1 cycle, followed by reassessment of Tumor Burden,
* If Tumor Burden classification is low after HDMP + Rituximab (lymph nodes < 5cm in diameter AND absolute lymphocyte count < 25k/uL), patients will initiate venetoclax dose ramp-up, with ramp-up schedule according to venetoclax package insert.
* Patients who still have a disease burden (lymphadenopathy > 5 cm or ALC > 25k/iL) that meets criteria for medium or high risk of TLS after 1 cycle of HDMP + Rituximab are given the option to repeat a 2nd cycle of HDMP + Rituximab prior to venetoclax dose ramp-up.

Upon completion of ramp-up (venetoclax to 400 mg), all patients will continue Venetoclax 400 mg (or highest tolerated dose) for up to 2 years. Patients will also continue rituximab 500 mg/m2 q 28 days through Cycle 6.

Endpoint Assessment:

1. Assessment of the disease burden after a maximum of 2 cycles of HDMP + Rituximab is the primary endpoint.
2. Assessment of the disease burden after 1 cycle of HDMP + Rituximab.
3. Assessment of the disease burden after 2 cycles of HDMP + Rituximab (for the subset of patients that do not meet criteria for low tumor burden after 1 cycle).
4. Clinical and laboratory TLS events between start of treatment and the completion of venetoclax dose-ramp up (Cycle 2, Day 1)
5. Presence or absence of detectable MRD in the marrow will be assessed after approximately 9 months of venetoclax and completion of treatment.
6. Radiology assessment after approximately 9 months of venetoclax and completion of study (unless prior imaging studies are without measurable disease)

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Subjects must be age 18 or older.
2. Both men and women of all races and ethnic groups are eligible for this trial.
3. Ability to understand and willingness to sign a written informed consent.
4. Diagnosis: CLL or SLL, as documented in the medical record
5. Disease Status/ Prior Therapy:

   * Must have had treatment for CLL/SLL with at least 1 line of prior therapy. (There is not requirement nor restriction for specific type of previous therapy, with the following exceptions: prior treatment with venetoclax within 6 months, prior progressive disease on venetoclax, or prior grade 3 or 4 toxicity (not including TLS) that directly lead to discontinuation of venetoclax; Prior HDMP/Rituximab is allowed unless there was no response (Stable Disease or Progressive Disease) or was within 3 months.)
   * Indication for CLL or SLL therapy based on international working group (iwCLL) guidelines, which include: constitutional symptoms, bulky or symptomatic lymphadenopathy, bulky or symptomatic splenomegaly, rapid doubling of the ALC (approximately 6 months or less), or Rai stage 3 or 4 disease.
   * Disease burden meets criteria for Medium or High Tumor Burden, based on Absolute lymphocyte count >/= 25k/uL or any lymph node 5 cm or greater in diameter. The ALC criteria must be met during the screening period. The imaging criteria may be based on radiologic study within 30 days of Cycle 0, Day 1.
6. Has recovered from the toxic effects of prior therapy to their clinical baseline.
7. Women of child-bearing potential (not postmenopausal for at least one year or not surgically incapable of bearing children) must agree to not become pregnant for the duration of the study. Both men and women must agree to use a barrier method of contraception for the duration of the study and until 5 half-lives after the final dose of venetoclax (approximately 1 week), and at least 5 half-lives of final dose of Rituximab.
8. ECOG performance status of 0-2
9. Adequate hematologic function: Platelet count >/= 30k/uL, hemoglobin > 7 g/dL, AND ANC > 500/uL. (Values may be lower if due to marrow infiltration by CLL).
10. Adequate renal function: creatinine clearance based on 24 hr collection >/= 40 ml/min; OR Calculated Creatinine clearance (CrCl) ≥ 40 mL/min (based upon the Cockcroft-Gault Equation [CrCl = (140-age) * actual wt (in kg) * (0.85 if female) / (72 * Cr)].
11. Adequate hepatic function:

    * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0X ULN
    * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Subject is known to be positive for HIV. (HIV testing is not required.)
2. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
3. Treatment with any of the following within 7 days prior to the first dose of venetoclax:

   * Steroid therapy for anti-neoplastic intent
   * moderate or strong cytochrome P450 3A (CYP3A) inhibitors (see Appendix C for examples)
   * moderate or strong CYP3A inducers (see Appendix C for examples)
4. Administration or consumption of any of the following within 3 days prior to the first dose of venetoclax:

   * grapefruit or grapefruit products
   * Seville oranges (including marmalade containing Seville oranges)
   * star fruit
5. Prior CLL therapy:

   * Biologic agent (monoclonal antibody) within 30 days for anti-neoplastic intent.
   * Chemotherapy (purine analog or alkylating agent) or target small molecule agent within 14 days or 5 half-lives (whichever is shorter), or has not recovered to less than CTC grade 2 clinically significant adverse effect(s)/toxicity(s) of previous therapy.
6. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
7. Known hypersensitivity to any of the study drugs
8. History of other malignancy that could affect compliance with the protocol or interpretation of results (example: patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are generally eligible. Patients with a malignancy that has been treated, but not with curative intent, will also be excluded, unless the malignancy has been in remission without treatment for 2 years prior to enrollment.)
9. Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds); or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks before the start of Cycle 0
10. Major surgery (within 4 weeks prior to the start of Cycle 0), other than for diagnosis
11. Women who are pregnant or lactating
12. Uncontrolled diabetes mellitus (related to high dose steroid risk)
13. Myocardial infarction within 6 months of starting study drug or other clinically significant heart disease (NYHA class 3 heart failure, uncontrolled hypertension)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2026-07-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Choi Michael, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study accrued four patients in total.
Pre-assignment Details: The the pre-planned sample size was 17.
Groups:
- Arm A: HDMP + rituximab as a means of debulking prior to initiating venetoclax.
  HDMP + rituximab as a means of debulking prior to initiating venetoclax.: - Patients will receive HDMP + Rituximab for 1 cycle, followed by reassessment of Tumor Burden,
  * If Tumor Burden classification is low after HDMP + Rituximab (lymph nodes < 5cm in diameter AND absolute lymphocyte count < 25k/uL), patients will initiate venetoclax dose ramp-up, with ramp-up schedule according to venetoclax package insert.
  * Patients who still have a disease burden (lymphadenopathy > 5 cm or ALC > 25k/iL) that meets criteria for medium or high risk of TLS after 1 cycle of HDMP + Rituximab are given the option to repeat a 2nd cycle of HDMP + Rituximab prior to venetoclax dose ramp-up.
Period: Overall Study
Arm/Group | Arm A
Started | 4
Completed | 2
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm A
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [66.75 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Prior Lines of Therapy [Median (Inter-Quartile Range); unit: Lines] | 1.5 [1 to 2.75]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Have a Decrease in Tumor Burden From Medium or High to Low
Description: Percentage of patients that have a decrease in tumor burden from levels of disease that meet "Medium/High-tumor burden" criteria to meet "Low tumor burden" criteria for disease burden following 1 or 2 cycles of HDMP + Rituximab.
  Low Tumor Burden = All measurable lymph nodes with the largest diameter < 5 cm by radiologic assessment AND ALC < 25k/uL
  Medium Tumor Burden = Any measurable lymph node with the largest diameter >/= 5 cm but < 10 cm by radiographic assessment OR ALC >/= 25k/uL
  High Tumor Burden = Any measurable lymph node with the largest diameter >/= 10 cm by radiologic assessment OR ALC >/= 25k/uL AND any measurable lymph node with the largest diameter >/= 5 cm
Time Frame: 28 or 56 days
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: Percentage of Patients That Have a Decrease in Tumor Burden From Medium to Low
Description: Percentage of patients that have a decrease in tumor burden from levels of disease that meet "Medium/High-tumor burden" criteria to meet "Low tumor burden" criteria for disease burden following 1 cycle of HDMP + Rituximab.
  Low Tumor Burden = All measurable lymph nodes with the largest diameter < 5 cm by radiologic assessment AND ALC < 25k/uL
  Medium Tumor Burden = Any measurable lymph node with the largest diameter >/= 5 cm but < 10 cm by radiographic assessment OR ALC >/= 25k/uL
Time Frame: 3 years
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Percentage of Patients That Have a Decrease in Tumor Burden if 2 Cycles of HDMP + Rituximab
Description: Percentage of patients that have a decrease in tumor burden from levels of disease that meet "Medium/High-tumor burden" criteria to meet "Low tumor burden" criteria for disease burden following 2 cycles of HDMP + Rituximab
  Low Tumor Burden = All measurable lymph nodes with the largest diameter < 5 cm by radiologic assessment AND ALC < 25k/uL
  Medium Tumor Burden = Any measurable lymph node with the largest diameter >/= 5 cm but < 10 cm by radiographic assessment OR ALC >/= 25k/uL
  High Tumor Burden = Any measurable lymph node with the largest diameter >/= 10 cm by radiologic assessment OR ALC >/= 25k/uL AND any measurable lymph node with the largest diameter >/= 5 cm
Time Frame: 56 days
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants | 2

4. Secondary Outcome: Rate of Laboratory TLS (Tumor Lysis Syndrome)
Description: Rate of laboratory TLS (from start of treatment until completion of venetoclax ramp-up)
Time Frame: 2.15 years
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Rate of Clinical TLS
Description: Rate of clinical TLS (from start of treatment until completion of venetoclax ramp-up)
Time Frame: 2.15 years
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Adverse Events by CTCAE4 Definitions
Description: Number of patients with non-hematological treatment-related adverse events by CTCAE4 definitions of grade 3 or higher, regardless of attribution
Time Frame: 2.15 years
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants
  Number of patients with non-hematological treatment-related adverse events of grade 3 or higher: Grade 3 or higher, related to treatment | 1
  Number of patients with non-hematological treatment-related adverse events of grade 3 or higher: < Grade 3, related or unrelated to treatment | 2
  Number of patients with non-hematological treatment-related adverse events of grade 3 or higher: No AEs | 1
  Number of patients with hematological treatment-related adverse events of grade 3 or higher: Grade 3 or higher, related to treatment | 0
  Number of patients with hematological treatment-related adverse events of grade 3 or higher: < Grade 3, related or unrelated to treatment | 3
  Number of patients with hematological treatment-related adverse events of grade 3 or higher: No AEs | 1

7. Secondary Outcome: Response Rates
Description: Overall Response rate, Partial Response rate, and Complete response rate per iwCLL criteria after 9 months of venetoclax and at completion of treatment
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 9 months and at end of study up to 3 years
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants
  Overall response rate around 9 months: Partial response | 0
  Overall response rate around 9 months: Complete response | 2
  Overall response rate around 9 months: Other | 2
  Overall response rate over the course of the study: Partial response | 1
  Overall response rate over the course of the study: Complete response | 2
  Overall response rate over the course of the study: Other | 1

8. Secondary Outcome: Undetectable Minimal Residual Disease (MRD) Rate
Description: Undetectable minimal residual disease (MRD) rate based on bone marrow biopsy after 9 months of venetoclax, and at completion of treatment
Time Frame: 3 years
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 4
Participants
  Undetectable MRD at 9 months: Undetectable MRD | 2
  Undetectable MRD at 9 months: Detectable | 2
  Overall response rate over the course of the study: Undetectable MRD | 3
  Overall response rate over the course of the study: Detectable | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm A
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=4)
Ear and Labyrinth disorders - other (Ear and labyrinth disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Edema limbs (General disorders) | 2 (2)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT04981912/Prot_SAP_000.pdf